CLINICAL TRIAL: NCT07262944
Title: Effect of Ultrasound-Guided External Oblique Intercostal Fascial Plane Block in Pediatric Patients Undergoing Otoplasty With Rib Cartilage Graft
Brief Title: EOI Block in Otoplasty With Rib Cartilage Graft
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Young-Eun Jang, professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2509-015-1674
Record Dates: First submitted 2025-11-13; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Postoperative Pain, Acute
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EOI block group (Experimental): Participants will receive ultrasound-guided external oblique intercostal (EOI) fascial plane block at the end of surgery. Under general anesthesia, a linear ultrasound probe (6-13 MHz) will be placed transversely at the 8th-9th intercostal space along the anterior axillary line. A 22-gauge, 50-80 mm needle will be advanced in-plane into the fascial plane between the external oblique and intercostal muscles, and 0.2% ropivacaine 0.5 mL/kg (maximum 30 mL) will be injected. Postoperative pain management will include intravenous patient-controlled analgesia (IV-PCA) with fentanyl.
  Interventions: Procedure: Ultrasound-guided External Oblique Intercostal (EOI) Fascial Plane Block
- Control group (No block) (Active Comparator): Participants will not receive the EOI block. All other perioperative management, including general anesthesia and postoperative intravenous patient-controlled analgesia (IV-PCA) with fentanyl, will be identical to the experimental group.
  Interventions: Procedure: Standard postoperative pain management (no EOI block)

INTERVENTIONS:
Procedure: Ultrasound-guided External Oblique Intercostal (EOI) Fascial Plane Block — Under general anesthesia, a linear ultrasound probe (6-13 MHz) is placed transversely at the 8th-9th intercostal space along the anterior axillary line. A 22-gauge, 50-80 mm needle is advanced in-plane into the fascial plane between the external oblique and intercostal muscles. After confirming correct needle placement, 0.2% ropivacaine 0.5 mL/kg (maximum 30 mL) is injected. The procedure is performed at the end of otoplasty with rib cartilage graft to provide postoperative analgesia.
  Arms: EOI block group
Procedure: Standard postoperative pain management (no EOI block) — Participants will not receive the EOI block. All other perioperative management, including general anesthesia and postoperative intravenous patient-controlled analgesia (IV-PCA) with fentanyl, will be identical to the experimental group.
  Arms: Control group (No block)

SUMMARY:
This randomized controlled trial aims to evaluate the effect of ultrasound-guided external oblique intercostal (EOI) fascial plane block on postoperative pain control and recovery in pediatric patients undergoing otoplasty with rib cartilage graft under general anesthesia. Participants aged 13 to 18 years will be randomly assigned to receive either EOI block with 0.2% ropivacaine or no block. Primary outcome is total opioid consumption within 24 hours after surgery. Secondary outcomes include NRS pain scores, incentive spirometry performance, incidence of atelectasis, and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* - Pediatric patients aged 13 to 18 years undergoing otoplasty with rib cartilage graft under general anesthesia at Seoul National University Children's Hospital
* Written informed consent obtained from parent or legal guardian, and assent from the patient

Exclusion Criteria:

* Unstable vital signs before surgery (heart rate <50 or >150 beats/min, systolic blood pressure <80 mmHg or >160 mmHg)
* Known hypersensitivity to ropivacaine or other amide-type local anesthetics
* Massive bleeding or shock
* Local infection at the injection site
* Sepsis
* History of allergy to opioid medications
* Severe renal dysfunction (creatinine >3.0 mg/dL)
* Severe hepatic dysfunction (AST or ALT >120 U/L)
* Any condition that, in the investigator's opinion, makes the subject unsuitable for study participation

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-12-01 (Estimated); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-08-30 (Estimated)

PRIMARY OUTCOMES:
Total opioid consumption within 24 hours after surgery | Within 24 hours after surgery
  Total amount of opioid analgesic (fentanyl) administered via intravenous patient-controlled analgesia (IV-PCA) and additional rescue doses within 24 hours postoperatively. The total dose will be normalized to body weight (µg/kg).

SECONDARY OUTCOMES:
Pain intensity at rest | Up to 24 hours after surgery
  Pain intensity at rest assessed using the Numerical Rating Scale (NRS, 0-10; higher scores = worse pain)
Pain intensity during deep breathing | Up to 24 hours after surgery
  Pain intensity during deep breathing assessed using the Numerical Rating Scale (NRS, 0-10; higher scores = worse pain)
Total non-opioid analgesic consumption | Up to 24 hours after surgery
  Total consumption of non-opioid analgesics (e.g., acetaminophen, NSAIDs) within 24 hours after surgery
Overall satisfaction with postoperative pain control | Up to 24 hours after surgery
  Overall patient satisfaction with postoperative pain control assessed using a 0-100 satisfaction scale (higher scores = better satisfaction)
Incidence of analgesic-related adverse events | Up to 24 hours after surgery
  Incidence of adverse events related to analgesics (nausea, vomiting, pruritus, dizziness, constipation, dry mouth, etc.)
Incentive spirometry performance | Within 30 minutes after PACU arrival
  Performance on incentive spirometry measured as the number of balls lifted at 30 minutes after PACU admission (Unit of Measure: number of balls (count))
Incidence of postoperative atelectasis | Up to 24 hours after surgery
  Presence or absence of atelectasis evaluated on chest X-ray approximately 24 hours postoperatively
Distribution of sensory block | At 30 minutes after PACU admission
  Dermatomal distribution of cold sensation loss assessed by alcohol swab test in the PACU by a blinded assessor, evaluated in standardized zones (midline, midclavicular, anterior/mid-axillary lines).
Sleep quality | Night of surgery
  Quality of sleep on the night of operation assessed on a 0-100 scale (0 = very poor, 100 = excellent).

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea